Abdominal hysterectomy and bilateral Magnesium sulfate infusion in oophorectomy surgery perioperative Study on "opioid consumption and its effect on postoperative analgesia

### **Data Collection Form**

| <b>DEMOGRA</b> | PHIC | DATA | ١: |
|----------------|------|------|----|
|----------------|------|------|----|

| | , |
|-------------------|-----------------------------------------|
| Name Surname | |
| Age | |
| Weight/Height/BMI | |
| Surgical Duration | |
| Anesthesia | |
| Duration | |
| BATON | |

#### INTRAOPERATIVE MONITORING;

| | Entranc | Induct | 5.min | 10 min | 15.min | 20.mi | 25 | 30 | 40 | 50.mi | 60.mi | 75 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | e | | | | | n | min | min | min | n | n | mi |
| | | 1 | | | | | | | | | | n |
| | | minut | | | | | | | | | | |
| | | e after | | | | | | | | | | |
| KH | | | | | | | | | | | | |
| OAB | | | | | | | | | | | | |
| SpO<br>2 | | | | | | | | | | | | |
| 2 | | | | | | | | | | | | |
| | 90 min. | 115 | 120.mi | 150.mi | 180.mi | | | | | | | |
| | | min | n | n | n | | | | | | | |
| KH | | | | | | | | | | | | |
| OAB | | | | | | | | | | | | |
| SpO | | | | | | | | | | | | |
| 2 | | | | | | | | | | | | |

### AT THE END OF SURGERY;

| Hypotensive requiring ephedrine episode number |
|------------------------------------------------|
| Bradycardia requiring atropine episode number |
| Total amount of remifentanil consumed |
| M.ALDRETE SCOR>8 arrival time in compilation |

## POSTOPERATIVE FOLLOW-UP;

| | | 30 min. | 2 H | 4.s | 6.s | 12.s | 24.s |
|---|---|---|---|---|---|---|---|
| Pain NRS | | | | | | | |
| | At rest: | | | | | | |
| | Active ( while coughing, | | | | | | |
| | walking ): | | | | | | |
| sedation | | | | | | | |
| Nausea-Vomiting | | | | | | | |

### AT THE END OF THE 24TH POSTOPERATIVE HOUR;

| first Tramadol request ( at what hour postoperatively |
|-------------------------------------------------------|
| was Tramadol administered) |
| Tramadol applications |
| Total amount of fentanyl consumed |

# 'Numerical Rating Scala'



## **Ramsay Sedation Scale**

| one: | Awake, restless and/or crying |
|------|--------------------------------------------------------------|
| 2: | Awake, calm, watching his surroundings |
| 3: | Sleepy but responds to verbal stimuli |
| 4: | Sleepy but glabellar responds immediately to tactile stimuli |
| 5: | Sleepy but glabellar responds slowly to tactile stimuli |
| 6: | Does not respond to warnings |

## Nausea-vomiting 'Verbal descriptive Scale '

| 0: | no nausea |
|------|-------------------|
| one: | mild nausea |
| 2: | moderate nausea |
| 3: | vomiting once |
| 4: | multiple vomiting |